CLINICAL TRIAL: NCT06304766
Title: Laparoscopic Versus Open Ablation of Liver Malignancies: a Randomized, Controlled Multicenter Trial
Brief Title: Open Versus Laparoscopic Ablation of Liver Malignancies
Acronym: OPTIMAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Hans-Christian Pommergaard, MD, DMSc, PhD, Clinical Research Associate Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-23015954
Record Dates: First submitted 2023-10-09; First posted 2024-03-12 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Hepatocellular Carcinoma; Cholangiocarcinoma; Liver Metastases
Keywords: Laparoscopic ablation; Open ablation; Complications; Ablation response; Quality of life; Randomized; Multicenter
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma

STUDY DESIGN:
Intervention Model Description: Approximately 80 patients will be randomized 1:1 between laparoscopic or open ablation after operability assesment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open ablation (Active Comparator): Laparotomy performed for open ablation of the tumor
  Interventions: Procedure: Open ablation
- Laparoscopic ablation (Experimental): Ablation of the tumor performed by laparoscopic approach
  Interventions: Procedure: Laparoscopic ablation

INTERVENTIONS:
Procedure: Laparoscopic ablation — Heat-based ablation modality performed by laparoscopy. Centers may use either radiofrequency or microwave ablation. The modality should be the same in both groups.
  Arms: Laparoscopic ablation
Procedure: Open ablation — Heat-based ablation modality performed by laparotomy. Centers may use either radiofrequency or microwave ablation. The modality should be the same in both groups.
  Arms: Open ablation

SUMMARY:
The purpose of this study is to compare laparoscopic ablation to open ablation of liver malignancies regarding complication rates and ablation response as well as quality of life following the surgery.

DETAILED DESCRIPTION:
Liver malignancies is a major cause of cancer-related mortality and the incidence is increasing. Patients with liver malignancies are often left with limited surgical treatment options due to extensive tumor burden or comorbidities. Ablation is a less invasive treatment for these patients that can be performed percutaneously, by laparoscopy or open surgery. Ablation during open surgery has a high potential of complications. Laparoscopic ablation presumably has a lower complication rate than during open surgery, yet still offers some of the same advantages needed for tumors in locations not favorable for percutaneous ablation. This study aims to compare laparoscopic ablation with ablation during open surgery to investigate a treatment option with a supposed lower complication rate and equally treatment effectiveness after one month.

ELIGIBILITY:
Inclusion Criteria:

* One or more tumors not amenable to percutaneous ablation, age ≥ 18, signed informed consent, diagnosis of primary liver cancer or liver metastases from any primary tumor, and tumor suitable for ablation as primary treatment.

Exclusion Criteria:

* Ablation performed in conjunction with resection, patients who cannot cooperate with the study, and patients who do not understand or speak Danish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Complications measured by the comprehensive complication index. | Complications are registered and clavien-dindo graded 30 days after surgery.
  Comprehensive Complication Index (CCI) scores compared between open and laparoscopic ablation groups. A higher CCI score represents a larger complication burden.

SECONDARY OUTCOMES:
Tumor ablation completeness. | 30 days after surgery.
  Presence of tumor remnants in ablation cavity one month after procedure evaluated with contrast enhanced CT.
Quality of Recovery score (QoR) | Before surgery and postoperative day 1, 7 and 30.
  Questionnaires are filled out prior to surgery and after
Quality of Life score (QoL) | Before surgery and on postoperative day 30.
  Questionnaires are filled out prior to surgery and after
Overall survival | Up to 90 days after surgery
  Overall and disease-free survival measured as survival status 90 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Christian Pommergaard, MD DMSc PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT06304766/Prot_SAP_000.pdf